CLINICAL TRIAL: NCT03685539
Title: Advanced CT Imaging Optimization for the Detection of Intracranial Metastasis
Brief Title: DECT in Imaging Patients With Solid Organ Cancer With Intracranial Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0303; NCI-2018-01984 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0303 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Malignant Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (DECT) (Experimental): Within 7 days before the standard Gamma Knife MRI, patients undergo DECT scan over 6 seconds at 1.5, 5, 10, and 20 minutes after receiving the contrast agent.
  Interventions: Procedure: Dual-Energy Computed Tomography

INTERVENTIONS:
Procedure: Dual-Energy Computed Tomography — Undergo DECT
  Other Names: DECT

SUMMARY:
This trial studies how well dual energy computed tomography (DECT) works in imaging patients with solid organ cancer that has spread to the brain. Imaging techniques, such as DECT, may help find and diagnose tumor cells and find out how far the tumor cells have spread in the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To optimize two major parameters of computed tomography (CT) imaging for optimal detection of intracranial metastatic lesions.

Ia. Virtual monochromatic image reconstruction. Ib. Contrast bolus timing. II. To measure the detection accuracy of CT compared to the diagnostic standard of care gadolinium-based "Gamma Knife (GK)" protocol magnetic resonance imaging (MRI).

OUTLINE:

Within 7 days before the standard Gamma Knife MRI, patients undergo DECT scan over 6 seconds at 1.5, 5, 10, and 20 minutes after receiving the contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with pathology-proven solid organ cancer
* MRI of the brain with contrast, positive for two or more metastatic lesions

  * One lesion with a single greatest diameter on contrast-enhanced MRI of 1 cm or greater
* Planned treatment with stereotactic radiosurgery

Exclusion Criteria:

* Known allergy to iodine-based contrast agents
* Patients with glomerular filtration rate (GFR) less than 30 or use of hemodialysis
* If prior nephrectomy, GFR less than 60
* Prior central nervous system malignancy
* Prior brain radiation
* Pregnant women are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Best diagnostic performance of computed tomography (CT) reconstruction parameters | Up to 2 years
  A repeated-measures analysis of variance with the Dunnett post hoc test will be used to determine the significance of the differences in the signal-to-noise (SNR) and contrast-to-noise (CNR) measurements at the optimal parameter setting, compared with all other parameter settings.
Accuracy of CT | Up to 2 years
  A Bland-Altman analysis will be used to show the agreement of number of lesions between optimal parametrized CT and the one of standard of care magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org